CLINICAL TRIAL: NCT05789862
Title: A Comprehensive Behavioral Health Evaluation and Intervention Program for Patients Undergoing Craniotomy for Brain Tumor
Brief Title: Behavioral Health Evaluation and Intervention Program for Patients Undergoing Craniotomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor portfolio adjustment
Sponsor: University of California, San Francisco (Other)
Collaborators: Clarity Squared Behavioral, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 211013; NCI-2023-02189 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Brain Tumor
Keywords: Health Technologies; Virtual Health Counseling; Quality of Life
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual behavioral health (Experimental): Participants will be assessed at 3 time points over the course the standard-of-care treatment before and after a scheduled craniotomy. At each time point, the participants will be asked to complete the questionnaires and engage in virtual counseling sessions.
  Interventions: Behavioral: Counseling Sessions; Behavioral: Quality of Life Questionnaires

INTERVENTIONS:
Behavioral: Counseling Sessions — Virtual sessions
  Other Names: Behavioral health counseling sessions
Behavioral: Quality of Life Questionnaires — Self administered questionnaires
  Other Names: Health related quality of life assessment (HRQoL)

SUMMARY:
This is a single center non-randomized, single-arm feasibility trial of the implementation of virtual behavioral health counseling sessions alongside standard-of-care treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of implementing behavioral health counseling sessions alongside standard of care treatment for brain tumor participants scheduled to undergo craniotomy for treatment.

SECONDARY OBJECTIVE:

I. To assess the acceptance of virtual behavioral health counseling sessions during the initial management of a newly diagnosed brain tumor.

II. To explore the rates of pre- and post-surgical mental health disorders in participants newly diagnosed with a brain tumor.

III. To explore pre- and post-surgical quality of life with virtual behavioral health counseling sessions during the initial management of a newly diagnosed brain tumor.

OUTLINE:

Participants will be given the opportunity to participate in virtual behavioral health counseling sessions at three time points relative to the scheduled tumor resection operation. All participants will receive questionnaires related to mental health, quality of life, and satisfaction with the study intervention. Participants who do not want to participate in the counseling sessions will be provided the option to complete the assessment tools related to mental health and quality of life only. Participants will be assessed over the course of 9 months related to standard-of-care treatment at the following time points: before the operation (baseline), 4 to 6 weeks following the operation, and 6 to 9 months following the operation. At each time point, the participants will fill out the questionnaires and engage in the virtual counseling sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years of age or older.
2. Able to understand study procedures and to comply with them for the entire length of the study.
3. Ability of individual or legal guardian/representative to understand a written informed consent document, and the willingness to sign it.
4. Documented diagnosis of a brain tumor.
5. PHQ-9 screening score of >= 5.
6. No prior surgical intervention, other than biopsy, for brain tumor.
7. Scheduled for craniotomy for brain tumor resection.

Exclusion Criteria:

1. Contraindication to any study-related procedure or assessment.
2. PHQ-9 scores of:

   1. < 5
   2. >= 20
   3. >= 1 point on Question number 9 - thoughts of self-harm or suicidality.
3. Require urgent or emergent surgical intervention or admission to the hospital prior to the scheduled surgery.
4. Prior surgical intervention for brain tumor.
5. Prior suicide attempt.
6. Prior hospitalization for psychiatric treatment.
7. Currently undergoing mental or behavioral health-related counseling or psychotherapy, other than currently taking an anti-depressant medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who completed program | Up to 9 months
  The proportion of enrolled patients that complete all three virtual behavioral health counseling sessions from time of study enrollment to the final behavioral health counseling session, approximately 6-9 months following the participants surgical operation, will be reported.

SECONDARY OUTCOMES:
Mean Client Satisfaction Questionnaire (CSQ-8) score | 6-9 months following surgery, approximately 1 day
  The CSQ-8 is an 8 item measure that will be utilized to measure the satisfaction with the behavioral telehealth counseling sessions. Items in the questionnaire are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction). Total scores range from 8 to 32, with higher scores indicating a greater satisfaction. The mean and standard deviation for each question and total questionnaire will be calculated and reported by group.
Mean Telehealth Usability Questionnaire (TUQ) score | 6-9 months following surgery, approximately 1 day
  The TUQ is a 21-question survey that was developed in response to the utilization of telehealth services in medical care. The survey is divided into 6 sections based on usefulness, ease-of-use, interface and interaction quality, reliability, satisfaction, and future use. Each question is scored on a 7-point Likert scale from 1 (Strongly Disagree) to 7 (Strongly Agree). The total score of each component is calculated by summing the item response scores in each component, with higher scores indicating a more positive experience with the intervention usability. The calculated mean and standard deviation by group will be reported.
Proportion of participants with a Patient Health Questionnaire 9 (PHQ-9) score >= 5 over time | Up to 9 months
  The PHQ-9 is used to measure depression symptoms. The total PHQ-9 score is calculated by combining the responses of the participant on questions addressing how bothered the participant has been by various problems over the past 2 weeks. Each of the 9 items is scored on a scale of 0 ("Not bothered at all") to 4 ("Nearly every day"). A total score of 5-9='Mild Depression Symptoms", 10-14="Minor Depression, Major Depression (mild), or Dysthymia", 15-19="Major Depression, moderately severe", and >20="Major Depression".
Mean score on the PHQ-9 over time | Up to 9 months
  The PHQ-9 is used to measure depression symptoms. The total PHQ-9 score is calculated by combining the responses of the participant on questions addressing how bothered the participant has been by various problems over the past 2 weeks. Each of the 9 items is scored on a scale of 0 ("Not bothered at all") to 4 ("Nearly every day"). A total score of 5-9='Mild Depression Symptoms", 10-14="Minor Depression, Major Depression (mild), or Dysthymia", 15-19="Major Depression, moderately severe", and >20="Major Depression". The PHQ-9 will be administered at Baseline, 4-6 weeks following surgery, and 6-9 months following surgery and the mean score and standard deviation will be reported.
Mean change in score on the on the PHQ-9 over time | Up to 9 months
  The overall mean change in score for each group on the PHQ-9 between the baseline visit and the second visit 4-6 weeks following surgery and the final follow-up visit, 6-9 months following surgery, will be reported.
Mean score on the General Anxiety Disorder-7 questionnaire (GAD-7) over time | Up to 9 months
  The GAD-7 is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater. The GAD-7 will be administered at Baseline, 4-6 weeks following surgery, and 6-9 months following surgery and the mean score and standard deviation will be reported.
Mean change in score on the on the GAD-7 over time | Up to 9 months
  The overall mean change in score for each group on the GAD-7 between the baseline visit and the second visit 4-6 weeks following surgery and the final follow-up visit, 6-9 months following surgery, will be reported.
Proportion of participants with at least 1 positive response on the Mini International Neuropsychiatric Inventory - Screen (M.I.N.I) over time | Up to 9 months
  The Mini International Neuropsychiatric Inventory - Screen (M.I.N.I) v7.0.2 is a brief, self-administered, structured interview designed to identify participants with positive responses for up to 19 adult behavioral disorders using Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria. A negative response to the screening questions usually means it is unlikely the participant has a major psychiatric disorder. A positive response to any questions in the M.I.N.I. Screen prompts the clinician to ask additional questions using the standard M.I.N.I. If a participant demonstrates a positive response, the M.I.N.I. Standard will be administered at that same time point. The M.I.N.I Screen will be administered at Baseline and 6-9 months following surgery
Proportion of participants with individual diagnoses on the M.I.N.I. Standard over time | Up to 9 months
  The M.I.N.I Standard is a full, clinician administered extended, structured interview which assesses the 17 most common disorders in mental health. The M.I.N.I. Standard will only be administered to participants with a positive response on the M.I.N.I Screen during the Baseline and 6-9 months following surgery assessments. Participants with negative responses at each assessment on the M.I.N.I Screen will not receive the M.I.N.I Standard at that assessment.
Mean score on the European Organisation For Research And Treatment Of Cancer Quality of Life Questionnaire, Brain (EORTC QLQ-BN20) over time | Up to 9 months
  The EORTC QLQ-BN20 consists of 20 questions; seven single item symptom scales (headaches, seizures, drowsiness, hair loss, itchy skin, leg weakness and bladder control), along with four multi-item scales (future uncertainty, visual disorder, motor dysfunction and communication deficit). Raw scores for the EORTC QLQ-BN20 items are computed by calculating the mean of the items in each subscale, or the item for each individual and linearly transform the scores to a 0-100 scale. A higher score represents worse QOL for all EORTC QLQ-BN20 scales and single items. The EORTC QLQ-BN20 will be administered at Baseline and 6-9 months following surgery
Mean change in score on the EORTC QLQ-BN20 over time | Up to 9 months
  The overall mean change in score for each group on the EORTC QLQ-BN20 between the baseline visit and final follow-up visit 6-9 months following surgery will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Hervey-Jumper, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No